CLINICAL TRIAL: NCT02957331
Title: Beta-Adrenergic Blockade for Suppression of Catecholamine Surge Following Traumatic Brain Injury: A Randomized Trial
Brief Title: Beta Blockade in in Traumatic Brain Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 15-04069-FB
Record Dates: First submitted 2016-10-31; First posted 2016-11-07 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2018-10

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol arm (Experimental): One half of qualifying and consenting subjects will be randomized to receive propranolol. This group will receive study drug 3 times daily (every 8 hours) starting at 20 mg. The dosage may be increased by up to 60 mg/day divided over three daily doses (or an additional 20 mg/dose) as necessary until the heart rate is less than 100. Study drug will be held for hypotension (systolic <100) or bradycardia (heart rate <60 beats per minute). The maximum daily dose for the treatment of hypertension of 640 mg will not be exceeded in this study.
  Interventions: Drug: Propranolol
- Non propranolol arm (No Intervention): Non beta blockade arm will receive standard of care treatment and will not receive beta blockade. If a subject randomized to no Inderal develops hypertension and increased heart rate, he/she will be treated according to standard of care by the trauma team caring for the patient.

INTERVENTIONS:
Drug: Propranolol
  Other Names: Inderal
  Arms: Propranolol arm

SUMMARY:
The purpose of this study is test the effect of beta-adrenergic blockade on mortality in patients with traumatic brain injury with the hypothesis being that the addition of beta blockade to the treatment regime of this patient population will lower mortality and supress the catecholamine surge that accompanies traumatic brain injury as compared to those who do not receive beta blockade.

Half the patients will be randomized to receive propranolol and half will be randomized to receive no beta blocker.

DETAILED DESCRIPTION:
The use of Beta-adrenergic blockade is not currently the standard of care of patients with traumatic brain injury. Traumatic brain injury is a common problem in our society with greater than 1.5 million cases occurring annually and over 50,000 deaths per year in the civilian population in the United States. Medical therapy has long consisted of monitoring intracranial pressure and supportive measures designed to limit intracranial pressure. Two retrospective observational studies completed at the University of Tennessee demonstrate that the addition of beta-adrenergic blockage to the treatment of the traumatic brain injury lessens mortality. The basis for conducting this study was established by retrospective data showing no harm to patients receiving Inderal and potential benefit. Available data, including data from the University of Tennessee, are retrospective and are limited to simple exposure to the drug. The proposed study will attempt to further quantify the effect by dosing with the drug to actual beta-blockade instead of simple exposure to the drug.

The effect of propranolol at the dosing levels used in this research will be determined by measurement of urinary catecholamines in both study arms and comparison of the actual effect of the drug on the catecholamine surge that occurs following traumatic brain injury will be determined.

Additionally, the effect of healthcare disparities on outcomes in patients with traumatic brain injury will be measured. Outcomes will be stratified by payer status and ethnicity to determine the effect each of these variables has on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 18 and older with isolated traumatic brain injury as defined by Glasgow Coma Scale score 12 or less with documented injury on head CT and limited injury to the rest of the body. (Abbreviated Injury Scale (AIS) must be < or = 3 from other body areas.)

Exclusion Criteria:

* Subjects <18 years of age, prisoners, those on beta-blockers as home medication, those who are pregnant, those with severe liver disease, those taking vasopressors, those with acute coronary syndrome, and those with severe injury to another body region (AIS >3).
* Subjects who cannot be enrolled within 48 hours of admission following acute resuscitation will not be enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Schroeppel, MD, Principal Investigator — University of Tennessee
Locations (1):
- Regional One Health, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kun LE, Gajjar A, Muhlbauer M, Heideman RL, Sanford R, Brenner M, Walter A, Langston J, Jenkins J, Facchini S. Stereotactic injection of herpes simplex thymidine kinase vector producer cells (PA317-G1Tk1SvNa.7) and intravenous ganciclovir for the treatment of progressive or recurrent primary supratentorial pediatric malignant brain tumors. Hum Gene Ther. 1995 Sep;6(9):1231-55. doi: 10.1089/hum.1995.6.9-1231. PMID 8527482
- [Background] Pople IK, Sanford RA, Muhlbauer MS. Clinical presentation and management of 100 infants with occipital plagiocephaly. Pediatr Neurosurg. 1996 Jul;25(1):1-6. doi: 10.1159/000121088. PMID 9055327
- [Background] Gajjar A, Sanford RA, Bhargava R, Heideman R, Walter A, Li Y, Langston JW, Jenkins JJ, Muhlbauer M, Boyett J, Kun LE. Medulloblastoma with brain stem involvement: the impact of gross total resection on outcome. Pediatr Neurosurg. 1996 Oct;25(4):182-7. doi: 10.1159/000121121. PMID 9293545
- [Background] Aggarwal R, Yeung D, Kumar P, Muhlbauer M, Kun LE. Efficacy and feasibility of stereotactic radiosurgery in the primary management of unfavorable pediatric ependymoma. Radiother Oncol. 1997 Jun;43(3):269-73. doi: 10.1016/s0167-8140(97)01926-9. PMID 9215786
- [Background] Chuba PJ, Aronin P, Bhambhani K, Eichenhorn M, Zamarano L, Cianci P, Muhlbauer M, Porter AT, Fontanesi J. Hyperbaric oxygen therapy for radiation-induced brain injury in children. Cancer. 1997 Nov 15;80(10):2005-12. doi: 10.1002/(sici)1097-0142(19971115)80:103.0.co;2-0. PMID 9366305
- [Background] Gajjar A, Sanford RA, Heideman R, Jenkins JJ, Walter A, Li Y, Langston JW, Muhlbauer M, Boyett JM, Kun LE. Low-grade astrocytoma: a decade of experience at St. Jude Children's Research Hospital. J Clin Oncol. 1997 Aug;15(8):2792-9. doi: 10.1200/JCO.1997.15.8.2792. PMID 9256121
- [Background] Muhlbauer M, Pfisterer W, Eyb R, Knosp E. Minimally invasive retroperitoneal approach for lumbar corpectomy and anterior reconstruction. Technical note. J Neurosurg. 2000 Jul;93(1 Suppl):161-7. doi: 10.3171/spi.2000.93.1.0161. PMID 10879777
- [Background] Fletcher DT, Warner WC, Muhlbauer MS, Merchant TE. Cervical subluxation after surgery and irradiation of childhood ependymoma. Pediatr Neurosurg. 2002 Apr;36(4):189-96. doi: 10.1159/000056056. PMID 12006754
- [Background] Williams RF, Magnotti LJ, Croce MA, Hargraves BB, Fischer PE, Schroeppel TJ, Zarzaur BL, Muhlbauer M, Timmons SD, Fabian TC. Impact of decompressive craniectomy on functional outcome after severe traumatic brain injury. J Trauma. 2009 Jun;66(6):1570-4; discussion 1574-6. doi: 10.1097/TA.0b013e3181a594c4. PMID 19509616
- [Background] DiCocco JM, Fabian TC, Emmett KP, Magnotti LJ, Zarzaur BL, Bate BG, Muhlbauer MS, Khan N, Kelly JM, Williams JS, Croce MA. Optimal outcomes for patients with blunt cerebrovascular injury (BCVI): tailoring treatment to the lesion. J Am Coll Surg. 2011 Apr;212(4):549-57; discussion 557-9. doi: 10.1016/j.jamcollsurg.2010.12.035. PMID 21463787
- [Background] Murphy RF, Cohen BH, Muhlbauer MS, Eubanks JW 3rd, Sawyer JR, Moisan A, Kelly DM. An accessory limb with lipomyelomeningocele in a male. Pediatr Surg Int. 2013 Jul;29(7):749-52. doi: 10.1007/s00383-013-3269-9. Epub 2013 Feb 8. PMID 23392915
- [Background] Klimo P Jr, Astur N, Gabrick K, Warner WC Jr, Muhlbauer MS. Occipitocervical fusion using a contoured rod and wire construct in children: a reappraisal of a vintage technique. J Neurosurg Pediatr. 2013 Feb;11(2):160-9. doi: 10.3171/2012.9.PEDS12214. Epub 2012 Nov 16. PMID 23157394
- [Background] Astur N, Klimo P Jr, Sawyer JR, Kelly DM, Muhlbauer MS, Warner WC Jr. Traumatic atlanto-occipital dislocation in children: evaluation, treatment, and outcomes. J Bone Joint Surg Am. 2013 Dec 18;95(24):e194(1-8). doi: 10.2106/JBJS.L.01295. PMID 24352780
- [Background] Astur N, Sawyer JR, Klimo P Jr, Kelly DM, Muhlbauer M, Warner WC Jr. Traumatic atlanto-occipital dislocation in children. J Am Acad Orthop Surg. 2014 May;22(5):274-82. doi: 10.5435/JAAOS-22-05-274. PMID 24788443
- [Background] Befeler AR, Gordon W, Khan N, Fernandez J, Muhlbauer MS, Sorenson JM. Results of delayed follow-up imaging in traumatic brain injury. J Neurosurg. 2016 Mar;124(3):703-9. doi: 10.3171/2015.4.JNS141257. Epub 2015 Oct 16. PMID 26473787

RESULTS

PARTICIPANT FLOW:
Groups:
- Propranolol Arm: One half of qualifying and consenting subjects will be randomized to receive propranolol. This group will receive study drug 3 times daily (every 8 hours) starting at 20 mg. The dosage may be increased by up to 60 mg/day divided over three daily doses (or an additional 20 mg/dose) as necessary until the heart rate is less than 100. Study drug will be held for hypotension (systolic <100) or bradycardia (heart rate <60 beats per minute). The maximum daily dose for the treatment of hypertension of 640 mg will not be exceeded in this study.
  Propranolol
Period: Overall Study
Arm/Group | Propranolol Arm | Non Propranolol Arm
Started | 14 | 12
Completed | 13 | 12
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol Arm | Non Propranolol Arm | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (19.0) | 53.0 (21.9) | 51.3 (20.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 9 | 7 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Mortality will be assessed at day 30 or at hospital discharge
Time Frame: 30 day
Measure: Number; unit: percentage of participants
Arm/Group | Propranolol Arm | Non Propranolol Arm
Number analyzed (Participants) | 13 | 12
percentage of participants | 7.7 | 33.3

2. Secondary Outcome: Urine Catecholamine Levels
Description: Urine catecholamine levels will be measured in the hospital laboratory
Time Frame: Collected at baseline, Day 2, Day 5, Day 10 and Day 14.
Measure: Least Squares Mean (Standard Error); unit: microgram/L
Arm/Group | Propranolol Arm | Non Propranolol Arm
Number analyzed (Participants) | 13 | 12
microgram/L
  Baseline | 236.4 (56.30) | 278.0 (52.1)
  Day 2 | 263.6 (51.56) | 181.9 (59.28)
  Day 5 | 308.5 (51.29) | 200.1 (48.19)
  Day 10 | 324.4 (51.67) | 216.7 (50.52)
  Day 14 | 375.3 (56.06) | 275.7 (44.06)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Propranolol Arm | Non Propranolol Arm
All-Cause Mortality (participants affected / at risk) | 1/13 | 4/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 1/13 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol Arm (N=13) | Non Propranolol Arm (N=12)
Tachycardia (Cardiac disorders) | 1 (1) | 0 — Rebound tachycardia occurred when propranolol was tapered off. A slower taper was used and this resolved the event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT02957331/Prot_SAP_000.pdf